CLINICAL TRIAL: NCT04868669
Title: In-home, Intensive Nutrition Counseling to Improve Gestational Weight Gain in Rural Bangladesh: A Cluster-Randomized Controlled Trial
Brief Title: Improving Maternal Nutrition in Matlab
Acronym: IMNiM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Obstetrical and Gynaecological Society of Bangladesh (OGSB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-19109
Record Dates: First submitted 2019-12-28; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Gestational Weight Gain
Keywords: nutrition counseling; gestational weight gain; cluster randomized controlled trial; birth weight
MeSH Terms: conditions — Gestational Weight Gain; Birth Weight

STUDY DESIGN:
Intervention Model Description: prospective, two-arm, parallel-group, equal allocation, open-label, community-based, cluster-randomized controlled trial
Masking Description: In this study, the blinding of the intervention is not feasible. However, the outcomes of the trial are objective in nature. Furthermore, the randomization and the statistical analysis will be carried out by someone unconnected to the allocation and enrollment process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In this arm, pregnant women, along with their influential family members such as mothers, mothers-in-law, and husbands, will receive monthly in-home, intensive nutrition counseling during the prenatal period.
  Interventions: Behavioral: In-home, intensive nutrition counseling
- Control (No Intervention): Pregnant women in this arm will receive standard antenatal care.

INTERVENTIONS:
Behavioral: In-home, intensive nutrition counseling — * Individualized sessions will be conducted by trained health workers following a standard document (counseling booklet)
  * The messages to be provided through the counseling will be contextualized
  * Sessions will start from the early second trimester and repeat monthly until 36 weeks of gestation
  * Counseling sessions will be conducted at the participant's place
  * Sessions will involve influential family members such as the husband, mother-in-law, mother, and the household head along with the pregnant women
  * Women will receive personalized feedback on their dietary intake pattern (dietary diversity) and the rate of weight gain in each session
  * Sessions will be tailored according to each participant's need and progress
  Arms: Intervention

SUMMARY:
Background: Maternal undernutrition and inadequate gestational weight gain (GWG) are prevalent in rural communities of low- and middle-income countries (LMICs). In Matlab, Bangladesh, 54% of the women fail to gain adequate weight (>4 kg) in the third trimester. Risks associated with inadequate GWG include giving birth to a small-for-gestational age (SGA) infant, low birth weight (LBW) infant, preterm birth (PTB), etc. Few contemporary studies examined the efficacy of nutrition counseling on GWG improvement in LMICs.

Objectives: The primary objective of this study is to assess whether in-home, intensive nutrition counseling during pregnancy, compared to standard antenatal care, could improve GWG among pregnant women in rural Bangladesh.

Methods: This prospective, two-arm, parallel group, equal allocation, open-label, community-based, cluster-randomized controlled trial will be conducted in the icddr,b service area of Matlab, a rural subdistrict of Bangladesh. Clusters will be randomly allocated 1:1 to the intervention arm in which pregnant women will receive monthly in-home, intensive nutrition counseling or the control arm in which pregnant women will receive standard antenatal care as offered by icddr,b and Govt. facilities. Fixed Site Clinics (FSCs) located at the homes of the community health research workers (CHRWs) will act as clusters. Of the 33 FSCs serving rural areas in the icddr,b service area, 20 will be selected randomly and listed. These 20 clinics will then be randomly allocated 1:1 to either an intervention or control group using a computer-generated random allocation sequence. To fulfil the required sample size, each selected CHRW will enroll 16 consecutive pregnancies. Required sample size is 16 women per cluster i.e. 160 women per arm. Eligible participants will be enrolled upon obtaining their consent by 13 and 6/7 weeks of gestation (first trimester) and followed up to 6 weeks postpartum. Trained health workers will visit the homes of the women in the intervention arm once a month and provide nutrition counseling to the women and her influential family members such as mothers, mothers-in-law and husbands. Both intention-to-treat and per-protocol analyses will be performed.

Outcome measures/variables: Proportion of women with inadequate rate of weight gain in the second and third trimester of pregnancy according to the US Institute of Medicine (IOM) 2009 guidelines is the primary outcome variable.

ELIGIBILITY:
Pregnant women permanently residing in the icddr,b service area of Matlab fulfilling the following criteria:

Inclusion Criteria:

* aged 18-39 years
* in the first trimester of pregnancy (before 14 weeks of gestation)
* BMI 16-24.99 kg/m^2 measured on enrollment
* willing to participate in the study

Exclusion criteria

* multiple pregnancy (carrying two or more fetuses)
* threatened abortion, persistent pervaginal bleeding, or cervical incompetence
* history of three or more consecutive abortions
* history of gestational diabetes, macrosomia, gestational hypertension, preeclampsia/eclampsia in a prior pregnancy
* chronic diseases, such as hypertension, heart disease, chronic obstructive pulmonary disease, chronic kidney disease, chronic liver disease, pancreatic diseases, Crohn's disease, ulcerative colitis, diabetes mellitus, thyroid dysfunction, immunological diseases, malignancy or any other diseases which could impede compliance with the study protocol
* taking medications known to influence fetal growth, such as insulin, thyroid hormones, glucocorticoids
* known case of serious psychiatric or behavioral disorders, such as schizophrenia, bipolar disorder
* scored as moderate or worse on enrollment on any one of the subscales of the Depression, Anxiety and Stress Scales-21 (DASS-21)
* inability to read or write Bengali
* belonging to moderately or severely food insecure households as measured by the Household Food Insecurity Access Scale (HFIAS)
* having a plan to move or deliver outside the study area
* women practicing some form of vegetarianism
* women belonging to a household from which another woman is already enrolled in the study

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This trial will focus on improving gestational weight gain in pregnant women. Hence, all the study participants are pregnant women.
Enrollment: 287 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
proportion of women with inadequate rate of weight gain in the second and third trimester of pregnancy according to IOM 2009 guidelines | Pre-delivery
  Pregnancy trimesters are defined as follows: 1st trimester (0 weeks - 13+6 weeks), 2nd trimester (14 completed weeks - 27+6 weeks), and 3rd trimester (28 completed weeks - childbirth). Rate of weight gain between two time points (trimesters) will be calculated by subtracting the weight measured at the first time point from the weight measured at the second time point and dividing the derived value by the difference in weeks between the two time points.

SECONDARY OUTCOMES:
total gestational weight gain (kg) | pre-delivery
rate of weight gain during the 2nd and 3rd trimester (kg/week) | pre-delivery
proportion of women with inadequate total GWG according to IOM criteria | pre-delivery
proportion of women with inadequate total GWG according to local criteria | pre-delivery
proportion of women with inadequate third trimester weight gain according to local criteria | pre-delivery
proportion of preterm births | at delivery
  childbirth before 37 completed weeks
maternal mid-upper arm circumference (MUAC) (mm) | baseline, 36 weeks of gestation, at delivery and 6 weeks post-partum
maternal weight (kg) | baseline, 36 weeks of gestation, pre-delivery, at delivery and 6 weeks post-partum
maternal body mass index (BMI) (kg/m^2) | baseline, 36 weeks of gestation, pre-delivery, at delivery and 6 weeks post-partum
  weight and height (at baseline) will be combined to report BMI
infant weight (g) | at birth (delivery) and after 4 weeks
infant length (cm) | at birth (delivery) and after 4 weeks
infant head circumference (cm) | at birth (delivery) and after 4 weeks
proportion of low birth weight (< 2500 g) infants | at birth (delivery)
proportion of small for gestational age (<10th percentile) infants according to Intergrowth-21st standards | at birth (delivery)
proportion of women with pregnancy complications e.g. anemia, preeclampsia | at delivery
proportion of women with obstetric complications e.g. induction of labor, caesarean section | at delivery
newborn Apgar score | at birth (delivery)
proportion of infants developing morbidity | 4 weeks after birth
proportion of infant mortality | 4 weeks after birth
dietary diversity score according to the "Guidelines for Measuring Household and Individual Dietary Diversity" | baseline, 36 weeks of gestation and 6 weeks post-partum
  score range: 0-9; higher scores indicate a better outcome
dietary diversity score according to the "Minimum Dietary Diversity for Women: A Guide to Measurement" | baseline, 36 weeks of gestation and 6 weeks post-partum
  score range: 0-10; higher scores indicate a better outcome
proportion of women with inadequate dietary diversity accroding to the "Minimum Dietary Diversity for Women: A Guide to Measurement" | baseline, 36 weeks of gestation and 6 weeks post-partum
  score range: 0-10; <5 indicates inadequate dietary diversity
energy consumption (kcal) | baseline, 36 weeks of gestation and 6 weeks post-partum
protein consumption (g) | baseline, 36 weeks of gestation and 6 weeks post-partum
proportion of women with symptoms of depression as measured by Depression, Anxiety, and Stress Scales-21 (DASS-21) scales | baseline, 36 weeks of gestation and 6 weeks post-partum
  DASS-21 is a validated, widely used, standardized self-report scale with 7 items in each subscale category of Depression, Anxiety, and Stress symptoms. Responses are scored on a 4-point Likert scale ranging from 0 (did not apply to me at all) to 3 (applied to me very much/most of the time), with higher scores indicating higher levels of depression, anxiety or stress.
proportion of women with symptoms of anxiety as measured by Depression, Anxiety, and Stress Scales-21 (DASS-21) scales | baseline, 36 weeks of gestation and 6 weeks post-partum
  DASS-21 is a validated, widely used, standardized self-report scale with 7 items in each subscale category of Depression, Anxiety, and Stress symptoms. Responses are scored on a 4-point Likert scale ranging from 0 (did not apply to me at all) to 3 (applied to me very much/most of the time), with higher scores indicating higher levels of depression, anxiety or stress.
proportion of women with symptoms of stress as measured by Depression, Anxiety, and Stress Scales-21 (DASS-21) scales | baseline, 36 weeks of gestation and 6 weeks post-partum
  DASS-21 is a validated, widely used, standardized self-report scale with 7 items in each subscale category of Depression, Anxiety, and Stress symptoms. Responses are scored on a 4-point Likert scale ranging from 0 (did not apply to me at all) to 3 (applied to me very much/most of the time), with higher scores indicating higher levels of depression, anxiety or stress.
healthcare seeking and services utilization e.g. number of prenatal visits | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: S. M. Tafsir Hasan, MBBS, MS, Principal Investigator — Nutrition and Clinical Services Division, icddr,b
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Chāndpur, Bangladesh

IPD SHARING:
Plan to Share IPD: No